CLINICAL TRIAL: NCT05867563
Title: A Phase I Clinical Trial Evaluating Tolerance, Safety, Pharmacokinetics, and Initial Effectiveness of TQB2103 for Injection in Patients With Advanced Cancers.
Brief Title: Clinical Trial Evaluating the Safety of the TQB2103 for Injection
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chia Tai Tianqing Pharmaceutical Group Nanjing Shunxin Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TQB2103-I-01
Record Dates: First submitted 2023-05-09; First posted 2023-05-22 (Actual); Last update posted 2023-07-10 (Actual); Status verified 2022-09

CONDITIONS: Advanced Malignant Neoplasm
MeSH Terms: interventions — Injections

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TQB2103 for Injection (Experimental): Dose escalation:
  intravenous infusion of TQB2103 for injection once every three weeks, 21 days as one treatment cycle.
  (0.5 mg/kg, 1.0 mg/kg, 2.0 mg/kg, 3.0 mg/kg, 4.0 mg/kg, 5.0mg/kg)
  Dose expansion:
  Chose one or two appropriate dose groups in the dose escalation experiment to expand.
  Interventions: Drug: TQB2103 for injection

INTERVENTIONS:
Drug: TQB2103 for injection — TQB2103 for injection is an antibody-drug conjugate targeting CLDN18.2. The drug structure mainly includes anti-humanized CLDN 18.2 antibody, linker and cytotoxic DDDXD, with Drug antibody Ratio (DAR) of 8.

SUMMARY:
TQB2103 injection is an antibody-drug conjugate (ADC) targeting claudin (CLDN) 18.2. This study aimed to evaluate the safety and tolerability, pharmacokinetic characteristics and immunogenicity of TQB2103 injection in patients with advanced malignant tumors as well as its initial effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* Patients with advanced malignant tumours confirmed by histology or cytology, disease progression or intolerance after adequate standard treatment, or lack of standard treatment options, or standard treatment is not applicable currently .
* Age: 18-75 years old; Eastern Cooperative Oncology Group Performance Status (ECOG PS) score: 0-1; The expected survival time is more than 3 months.
* Patients who can provide fresh-collected or stored tumour tissue samples within 2 years for Claudin 18.2 expression level detection were preferentially enrolled, and those who cannot provide samples during the dose-escalation stage were also eligible to participate in the study; In the dose-expansion stage, subjects who could not provide tumour tissue samples for Claudin 18.2 expression level detection needed to be discussed with the investigators on a case-by-case basis, and enrollment may be allowed according to the specific situation.
* At least one evaluable tumour lesion according to Response Evaluation Criteria In Solid Tumors (RECIST) v1.1 in the dose-escalation study and at least one measurable lesion in the dose-expansion study (the lesion that received radiotherapy can be used as the target lesion after definite progression according to RECIST v1.1 evaluation).
* Good function of major organs.
* Fertile subjects should agree that contraception must be used during the study and for 6 months after the end of the study; Women of childbearing age had a negative serum pregnancy test within 7 days prior to study enrollment and had to be non-lactating subjects.
* Evidence of a personally signed and dated informed consent document indicating that the patient has been informed of all pertinent aspects of the study.

Exclusion Criteria:

* Comorbidities and medical history:

  1. Have developed or are currently concurrent with other malignant tumors within the past 5 years.
  2. Have a high risk of Gastrointestinal (GI) bleeding, or have active severe GI disease.
  3. Patients with current interstitial lung disease or pulmonary fibrosis, pneumoconiosis, radiation pneumonitis, severe impairment of lung function, etc., which may interfere with the detection and management of suspected drug-related pulmonary toxicity.
  4. All reversible adverse events caused by any previous treatment have not recovered to CTCAE 5.0 grade ≤ grade 1, before the first dose of the investigational drug.
  5. Major surgical treatment, open biopsy, or significant traumatic injury within 4 weeks before the start of study treatment; Elective surgery was required during the trial; Or have wounds, ulcers or fractures that have not healed for a long time.
  6. Occurrence of arterial/venous thrombosis events within 6 months, such as cerebrovascular accident, deep vein thrombosis, and pulmonary embolism; People who have a history of psychotropic drug abuse and cannot abstain from it or have mental disorders.
  7. Subjects with any severe and/or uncontrolled illness.
* Cancer-related symptoms and treatment:

  1. Received systemic antineoplastic therapy such as radical surgery, chemotherapy, radical radiotherapy or immunotherapy, biological therapy or participated in Clinical trials of other interventional antineoplastic drugs within 4 weeks before the initiation of study treatment.
  2. Prior therapy against the Claudin18.2 target, such as Claudin18.2 monoclonal antibodies, bispecific antibody, ADC, or chimeric antigen receptor T-cell immunotherapy (CAR-T).
  3. Tumour has invaded important blood vessels on imaging (Computed Tomography (CT) or Magnetic Resonance Imaging(MRI)) or judged by the investigator to be highly likely to invade important blood vessels during the follow-up study.
  4. Poorly controlled pleural, pericardial or peritoneal effusion requiring repeated drainage, judged by the investigator to be unsuitable for enrollment.
  5. Subjects with known active central nervous system metastases and/or meningeal metastases or spinal cord compression.
* Study treatment-related:

  1. A history of vaccination with the live attenuated vaccine within 28 days before initiation of study treatment or a planned vaccination with live attenuated vaccine during the study.
  2. The subject has a history of severe hypersensitivity after previous exposure to a humanized monoclonal antibody or acute or delayed hypersensitivity or intolerance to known components of TQB2103.
  3. Requiring systemic therapy within 2 years before initiation of study treatment.
* Subjects with concomitant diseases that seriously endanger the safety of the subjects or affect the completion of the study, or subjects who are considered to be unsuitable for enrollment for other reasons, according to the judgment of the investigators.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Estimated)
Dates: Start 2023-07-04 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicity (DLT) | During the first treatment cycle (21 days).
  DLT was defined as toxicities that meet pre-defined severity criteria according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v5.0, and assessed as having suspected relationship to investigational drug that occurred within the first treatment cycle (21 days).
Maximum tolerated dose (MTD) | During the first treatment cycle (21 days).
  MTD was defined as the highest dose at which dose limiting toxicity (DLT) occurred in less than 33% of patients.
Recommended Phase II Dose (RP2D) | During the first treatment cycle (21 days).
  The RP2D of anticancer agents is determined traditionally by dose-limiting toxicities. Nontoxicity or biological endpoints such as pharmacokinetics, pharmacodynamics, and efficacy can also be used to identify RP2D.

SECONDARY OUTCOMES:
The area under the curve (AUC) | 2 hours pre-dose, 0, 2, 4, 7, 24, 72, 144, 312, 504 hours (when necessary) after dose on cycle 1 and cycle 3; 2 hours pre-dose, 0 hour, 504 hours (when necessary) after dose on cycle 2, cycle 4, cycle 6, cycle 8. Each cycle is 21 days.
  The area under the curve (AUC) of serum or plasma concentration of ADC drug, total antibody, and small molecule toxin.
Peak concentration (Cmax) | 2 hours pre-dose, 0, 2, 4, 7, 24, 72, 144, 312, 504 hours (when necessary) after dose on cycle 1 and cycle 3; 2 hours pre-dose, 0 hour, 504 hours (when necessary) after dose on cycle 2, cycle 4, cycle 6, cycle 8. Each cycle is 21 days.
  Maximum observed concentration (Cmax) of ADC drug, total antibody and small molecule toxin after administration.
Immunogenicity | 120 minutes pre-dose on Cycle 1 Day 1, Cycle 2 Day1, Cycle 4 Day1, Cycle 7 Day1, Cycle 12 Day1; 90 days after the last infusion. Each cycle is 21 days.
  Incidence of anti-drug antibody (ADA)
Terminal half-life (T1/2) | 2 hours pre-dose, 0, 2, 4, 7, 24, 72, 144, 312, 504 hours (when necessary) after dose on cycle 1 and cycle 3; 2 hours pre-dose, 0 hour, 504 hours (when necessary) after dose on cycle 2, cycle 4, cycle 6, cycle 8. Each cycle is 21 days.
  T1/2 is the time required to decrease the concentration of a drug within the body by one-half.
Apparent Clearance (CL/F) | 2 hours pre-dose, 0, 2, 4, 7, 24, 72, 144, 312, 504 hours (when necessary) after dose on cycle 1 and cycle 3; 2 hours pre-dose, 0 hour, 504 hours (when necessary) after dose on cycle 2, cycle 4, cycle 6, cycle 8. Each cycle is 21 days.
  Apparent clearance refers to the rate of drug removal in the body, which reflects the degree of drug elimination in the body, as well as the bioavailability of the drug in the body.
Apparent distribution volume (Vss/F) | 2 hours pre-dose, 0, 2, 4, 7, 24, 72, 144, 312, 504 hours (when necessary) after dose on cycle 1 and cycle 3; 2 hours pre-dose, 0 hour, 504 hours (when necessary) after dose on cycle 2, cycle 4, cycle 6, cycle 8. Each cycle is 21 days.
  When the drug distribution in plasma and tissue reaches equilibrium, the required body fluid volume for drug distribution in the body according to the plasma drug concentration at this time.
Objective Response Rate (ORR) | Up to 2 years
  Defined as the percentage of complete response (CR) and partial response (PR) assessed by Response Evaluation Criteria In Solid Tumors (RECIST) v1.1 criteria.
Disease control rate (DCR) | Up to 2 years
  Defined as the proportion of subjects with CR, PR, or stable disease (SD).
Duration of Response (DOR) | Up to 2 years
  Defined as the time from first documented response to documented disease progression.
Progress Free Survival (PFS) | Up to 2 years
  Defined as the time from the first dose of TQB2103 to the first occurrence of disease progression or death from any cause.
Overall Survival (OS) | Up to 2 years
  Overall survival refers to the time from the first treatment to death from any cause.
Adverse event rate | Up to 2 years
  The occurrence of all adverse events (AEs), serious adverse events (SAEs) and treatment-related adverse events (TEAEs) evaluated by Common Terminology Criteria for Adverse Events (CTCAE) 5.0.

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Hunan Cancer Hospital, Changsha, Hunan
  - Xuzhou Central Hospital, Xuzhou, Jiangsu
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No